CLINICAL TRIAL: NCT05291754
Title: 3D Printed PEEK Implants for Cranioplasty
Acronym: PEEKCP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Region Skane (Other); Lund University (Other)
Responsible Party: Principal Investigator, Peter Siesjö, Professor, Skane University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ver1.2
Record Dates: First submitted 2021-11-26; First posted 2022-03-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Skull Defect
Keywords: PEEK; Cranioplasty; 3D printer

STUDY DESIGN:
Intervention Model Description: Prospective, non randomised and single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cranioplasty PEEK (Other)
  Interventions: Device: PEEK Cranioplasty

INTERVENTIONS:
Device: PEEK Cranioplasty — 3D printed PEEK skull implant

SUMMARY:
This study is a non-randomised and single center study with patients needing an artificial skull bone eg cranioplasty. 40 patients will be implanted with in house manufactured polyether ether ketone (PEEK) implants using a fused filament fabrication 3D printer. The primary aim is to ascertain safety and feasibility of the procedure. The secondary aim is to compare complication rates with conventional methods such as autologous bone and polymethylmetacrylate (PMMA).

DETAILED DESCRIPTION:
Cranioplasty is the surgical repair of a congenital or cranial defects after head trauma, infection or decompressive craniectomy. Although some patients can tolerate cranial defects for varied periods of time, cranioplasty is mostly indicated due to the increased risk of additional brain trauma, local pain or impaired CSF circulation but also aesthetic and psychological issues. The gold standard for repair since many years is cranioplasty with autologous bones . However, sometimes it not feasible to use the patient's autologous bone due to infections, trauma, bone graft resorption and donor-site morbidity. To replace the autologous bone grafts several different materials have been used, or are in use, as titanium meshes, hydroxyapatite cement and plastic resins as polymethyl methacrylate (PMMA) and porous polyethylene. Some of these have gathered increased interest due to advancements in technology for manufacture of these materials, and also the possibility to create custom made implants or moulds.

The present study aims to assay safety and feasibility of in house 3D printed medical grade PEEK implants in research persons with acquired skull defects.

The implants will be manufactured after 3D rendering from CT images of the skull defects, sterilised and aseptically inserted in the defects by means of a surgical intervention.

A safety interim analysis will be performed after inclusion of 10 patients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for cranioplasty
* Informed consent

Exclusion Criteria:

* No informed consent
* Implant size greater than 12x12 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2025-12-26 (Actual); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Performed PEEK implants | At end of surgical procedure, up to 2 months after inclusion
  Percentage of performed PEEK implants out of included patients.
Safety of PEEK implants | 1 year
  Survival percentage of PEEK implants. Will be compared to historical PMMA and autologous bone implants.

SECONDARY OUTCOMES:
Exposure time of PEEK implants compared to PMMA implants. | During surgical procedure, up to 2 months after inclusion.
  Compare exposure time for PEEK implant during surgery with historical PMMA implants made in 3D printed mold.
Complications of PEEK implants | 12 months
  Complications after PEEK implants other than those leading to extraction of implant will be compared to historical PMMA and autologous bone implants.

CONTACTS AND LOCATIONS:
Overall Officials: Einar Heiberg, MD, PhD, Study Director — Skane University Hospital
Locations (1):
- Department of Neurosurgery, Lund, Sweden